CLINICAL TRIAL: NCT04208178
Title: EPIK-B2: A Two Part, Phase III, Multicenter, Randomized (1:1), Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of Alpelisib (BYL719) in Combination With Trastuzumab and Pertuzumab as Maintenance Therapy in Patients With HER2-positive Advanced Breast Cancer With a PIK3CA Mutation
Brief Title: Study of Alpelisib (BYL719) in Combination With Trastuzumab and Pertuzumab as Maintenance Therapy in Patients With HER2-positive Advanced Breast Cancer With a PIK3CA Mutation
Acronym: EPIK-B2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBYL719G12301; 2024-512050-13-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2019-12-12; First posted 2019-12-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Advanced HER2+Breast Cancer
Keywords: BYL719; alpelisib; Advance Breast Cancer; maintenance; HER2 positive; induction; PI3K; Trastuzumab; Pertuzumab
MeSH Terms: interventions — Alpelisib; Trastuzumab; pertuzumab

STUDY DESIGN:
Intervention Model Description: Part 1 was the open-label, safety run-in part of the study designed to confirm the recommended phase 3 dose (RP3D) dose of alpelisib in combination with trastuzumab and pertuzumab. Following Part 1, Part 2 was initiated, which is the randomized, Phase III part of the study with two treatment arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 was the open-label, safety run-in part of the study designed to confirm the recommended phase 3 dose (RP3D) dose of alpelisib in combination with trastuzumab and pertuzumab. Once the alpelisib dose was confirmed, Part 2 with masking for participant, care provider, investigator and outcome assessor started. Participants in Part 2 are to be unblinded with the implementation of protocol amendment 03.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Alpelisib + Trastuzumab + Pertuzumab (Experimental): In the Part 1, up to 3 alpelisib dose levels may be sequentially tested in 3 cohorts of subjects:
  Cohort A: Alpelisib 300mg + trastuzumab (6mg/kg) + pertuzumab (420 mg) Cohort B: Alpelisib 250 mg+ trastuzumab (6mg/kg) + pertuzumab (420 mg) Cohort C: Alpelisib 200mg + trastuzumab (6mg/kg) + pertuzumab (420 mg)
  Interventions: Drug: Alpelisib; Drug: Trastuzumab; Drug: Pertuzumab
- Part 2: Alpelisib + Trastuzumab + Pertuzumab (Experimental): Trastuzumab (6mg/kg) + pertuzumab (420 mg) in combination with 200mg alpelisib, with potential for intra-participant dose escalation to 250 mg
  Interventions: Drug: Alpelisib; Drug: Trastuzumab; Drug: Pertuzumab
- Part 2: Alpelisib matching Placebo + Trastuzumab + Pertuzumab (Placebo Comparator): Trastuzumab (6mg/kg) + pertuzumab (420 mg) in combination with 200 mg alpelisib matching placebo, with potential for intra-participant dose escalation to 250 mg
  Interventions: Drug: Alpelisib matching Placebo; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Alpelisib — Alpelisib orally taken - continuous once daily, in a 21-day cycle.
  Other Names: BYL719
  Arms: Part 1: Alpelisib + Trastuzumab + Pertuzumab; Part 2: Alpelisib + Trastuzumab + Pertuzumab
Drug: Alpelisib matching Placebo — Alpelisib matching placebo orally taken - continuous once daily, in a 21-day cycle
  Arms: Part 2: Alpelisib matching Placebo + Trastuzumab + Pertuzumab
Drug: Trastuzumab — Trastuzumab 6mg/kg given intravenously - Day 1 of Cycle 1, and on Day 1 of every cycle thereafter (Cycle=21 days)
Drug: Pertuzumab — Pertuzumab 420 mg given intravenously - Day 1 of Cycle 1, and on Day 1 of every cycle thereafter (Cycle=21 days)

SUMMARY:
The purpose of this two part multicenter, randomized, double-blind, placebo-controlled, Phase III study is to evaluate the efficacy and safety of alpelisib compared to alpelisib matching-placebo in combination with trastuzumab and pertuzumab as maintenance treatment of patients with HER2-positive advanced breast cancer whose tumor harbors a PIK3CA mutation following induction therapy with a taxane in combination with trastuzumab and pertuzumab. Part 1 is the open-label, safety run-in part of the study, designed to confirm the recommended phase 3 dose (RP3D) dose of alpelisib in combination with trastuzumab and pertuzumab. Following Part 1, Part 2 will be initiated, which is the randomized, Phase III part of the study.

DETAILED DESCRIPTION:
The recruitment for this study was permanently halted as of 07-Dec-2022 with the intent of ending the study early because of the evolving treatment landscape and changing paradigms for HER-2 positive BC therapy. This decision was not triggered by any new or unexpected safety findings. Participants in Part 1 will be allowed to continue study treatment (alpelisib in combination with trastuzumab and pertuzumab) if they are deriving clinical benefit as assessed by the investigator and after discussion with the participant and documentation in the medical record. All participants in Part 2 will be unblinded for knowledge of treatment allocation and continuity treatment planning.Participants in the experimental arm will be allowed to continue alpelisib in combination with trastuzumab and pertuzumab based on investigator's judgement and benefit/risk assessment.Participants in Part 2 who are still receiving study treatment in the control arm with alpelisib matching-placebo will not be allowed cross-over to the experimental arm. These participants will be allowed to continue on trastuzumab and pertuzumab if they are deriving clinical benefit as assessed by the investigator and after discussion with the participant and documentation in the medical record.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically-confirmed HER2-positive breast cancer that is advanced (loco-regionally not amenable to surgery or is metastatic).
* Participant has received pre-study induction therapy with up to and including a maximum of 8 cycles of a taxane (docetaxel, paclitaxel, or nab-paclitaxel), plus trastuzumab and pertuzumab. 4 or 5 cycles of induction therapy are permitted if discontinuation of taxane was due to taxane toxicity. Of note, participants enrolled in Part 1 of this study received 4-6 cycles of pre-study induction therapy.
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Participant has adequate bone marrow and organ function
* Applies only to Part 2: Participant has a PIK3CA mutation(s) present in tumor prior to enrollment, locally confirmed per test listed in protocol or as determined by a Novartis designated central laboratory.

Exclusion Criteria:

* Participant with inflammatory breast cancer at screening.
* Participant with evidence of disease progression during the pre-study induction therapy and prior to first dose of alpelisib (or alpelisib/alpelisib matching-placebo for Part 2)
* Participant with an established diagnosis of diabetes mellitus type I or uncontrolled type II based on fasting plasma glucose (FPG) and HbA1c.
* Participant has a known history of acute pancreatitis within 1 year of screening or past medical history of chronic pancreatitis
* Participant has clinically significant, uncontrolled heart disease and/or recent cardiac events
* Participant has a history of Steven-Johnson Syndrome (SJS), erythema multiforme (EM) or Toxic Epidermal Necrolysis (TEN).
* Participant has currently documented pneumonitis/interstitial lung disease

Other protocol-defined Inclusion/Exclusion may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
Part 1: Incidence of dose limiting toxicities (DLTs) for each dose level | 6 weeks
  Incidence of DLTs during the first 6 weeks of treatment for each dose level associated with administration of alpelisib in combination with trastuzumab and pertuzumab
Part 2: Progression Free Survival (PFS) | Up to approximately 38 months
  PFS is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause. PFS is based on local investigator assessment and using RECIST 1.1 criteria

SECONDARY OUTCOMES:
Part 1: Alpelisib concentrations by timepoint and dose level | Day 8 of Cycle 1 and then Day 1 of Cycle 2, Cycle 4, Cycle 6 and Cycle 10 (Cycle = 21 days)
  Characterize exposure of alpelisib when administered in combination with trastuzumab and pertuzumab
Part 2: Overall survival (OS) (Key Secondary) | Up to approximately 70 months
  OS is defined as the time from date of randomization to date of death due to any cause
Part 2: Summary statistics of alpelisib concentrations by timepoint and dose level | Day 8 of Cycle 1 and then Day 1 of Cycle 2, Cycle 4, Cycle 6 and Cycle 10 (Cycle = 21 days)
  Characterize exposure of alpelisib when administered in combination with trastuzumab and pertuzumab
Part 2: Overall response rate (ORR) with confirmed response | Up to approximately 38 months
  ORR is defined as the percentage of patients with best overall response of complete response (CR) or partial response (PR) based on local investigator's assessment according to RECIST 1.1.
Part 2: Clinical Benefit Rate (CBR) with confirmed response | Up to approximately 38 months
  Clinical benefit rate is defined as the percentage of patients with a best overall response of complete response (CR) or partial response (PR) or Stable disease (SD) or Non-CR/Non-progressive disease (PD) lasting more than 24 weeks based on local investigator assessment.
Part 2: Time to response (TTR) based on local radiology assessments | Up to approximately 38 months
  Time to response (TTR) is defined as the time from the date of randomization to the first documented response of either complete response (CR) or partial response (PR), which must be subsequently confirmed (although date of initial response is used, not date of confirmation). TTR will be assessed using RESIST 1.1 criteria.
Part 2: Duration of response (DOR) with confirmed response | Up to approximately 38 months
  DOR is calculated as the time from the date of first documented response (complete response (CR) or partial response (PR)) to the first documented date of progression or death due to underlying cancer.
Part 2: Change in Functional Assessment of Cancer Therapy - Breast (FACT-B) treatment outcomes index (TOI) from baseline | Baseline, up to approximately 38 months
  The FACT-B is a 37-item instrument designed to measure five domains of Health-Related Quality of Life (HRQOL) in breast cancer patients: Physical Well-being (PWB), Social/family Well-being (SWB), Emotional Well-being (EWB), Functional Well-being (FWB) as well as a Breast Cancer Subscale (BCS).
  The FACT-B TOI is a composite of PWB, FWB and BCS scores. Total score ranges from 0 to 96. Higher FACT-B TOI scores represent better QoL.
  Change from baseline in FACT-B TOI scores will be calculated
Part 2: Time to deterioration in FACT-B TOI (defined as a ≥ 5 point decrease from baseline) | Baseline, up to approximately 38 months
  The FACT-B is a 37-item instrument designed to measure five domains of Health-Related Quality of Life (HRQOL) in breast cancer patients: Physical Well-being (PWB), Social/family Well-being (SWB), Emotional Well-being (EWB), Functional Well-being (FWB) as well as a Breast Cancer Subscale (BCS).
  The FACT-B TOI is a composite of PWB, FWB and BCS scores. Total score ranges from 0 to 96. Higher FACT-B TOI scores represent better QoL. Definitive deterioration is defined as the time from the date of randomization to the date of event defined as at least 5-point worsening from baseline with no later improvement above this threshold observed during the course of the treatment or until death due to any cause in FACT-B TOI score
Part 2: PFS based on local radiology assessments by PIK3CA mutation status | Up to approximately 38 months
  Evaluate the association between PIK3CA mutation status as measured in ctDNA at baseline with PFS upon treatment with alpelisib. PFS will be assessed using RECIST 1.1 criteria for patients by PIK3CA mutation status assessed in ctDNA at baseline.
Part 2: Time to definitive deterioration of Eastern Cooperative Group of Oncology Group (ECOG) performance status | Baseline, up to approximately 38 months
  ECOG: participant's performance status was measured on a 6-point scale: 0= fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light and sedentary nature; 2= ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50 percent (%) of waking hours; 3= capable of only limited self-care, confined to bed/chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed/chair: 5= dead. Time to definitive deterioration in ECOG PS is defined as the time from the date of randomization to the date when the ECOG PS has definitely deteriorated by at least one category compared with baseline. Deterioration is considered definitive if there is no subsequent improvement in ECOG PS back to baseline category or above.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (2):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of California LA, Los Angeles, California
- Belgium (2):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- China (2):
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shanghai
- France (2):
  - Novartis Investigative Site, Saint-Cloud, Hauts De Seine
  - Novartis Investigative Site, Saint-Herblain
- Novartis Investigative Site, Florence, FI, Italy
- Novartis Investigative Site, Kuala Lumpur, Malaysia
- Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com